CLINICAL TRIAL: NCT05697016
Title: Sivelestat for the Treatment of Adult Patients With Acute Respiratory Distress Syndrome Due to COVID-19: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Sivelestat for Acute Respiratory Distress Syndrome Due to COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Guangzhi Shi, Doctor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HX-B-2022083
Record Dates: First submitted 2023-01-16; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Respiratory Infection Virus; Respiratory Failure
Keywords: ARDS; COVID-19; Sivelestat; Randomized Trial
MeSH Terms: conditions — Respiratory Insufficiency; COVID-19 | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Sivelestat group (Experimental): The patients in this group will receive sivelestat sodium via continuous intravenous infusion (0.2mg/kg/h) over a 24-hour period for 7 days
  Interventions: Drug: Sivelestat Sodium for Injection
- The Placebo group (Placebo Comparator): The patients in this group will receive the placebo via continuous intravenous infusion (0.2mg/kg/h) over a 24-hour period for 7 days
  Interventions: Drug: The Placebo

INTERVENTIONS:
Drug: Sivelestat Sodium for Injection — Sivelestat, a specific inhibitor of neutrophil elastase; sodium N-[2-[4-(2,2-dimethylpropionyloxy) phenyl-sulfonylaminobenzoyl]amino-acetate tetrahydrate]
  Other Names: Supportive management of ARDS (e.g., protective ventilation strategy, prone positioning and/or VV-ECMO, etc.) based on currently recommended practice guidelines
  Arms: the Sivelestat group
Drug: The Placebo — Excipients used for the sivelestat sodium
  Other Names: Supportive management of ARDS (e.g., protective ventilation strategy, prone positioning and/or VV-ECMO, etc.) based on currently recommended practice guidelines
  Arms: The Placebo group

SUMMARY:
A randomized, double-Blind, placebo-controlled trial aimed to investigate the safety and efficacy of sivelestat on treating adult patients with COVID-19-related acute respiratory distress syndrome (ARDS)

DETAILED DESCRIPTION:
This study is designed as a randomized, double-blind, placebo-controlled clinical trial, and is planned to be conducted at 3 clinical centers in China from January 1, 2023, to January 31, 2024. During the study period, we intend to enroll a total of 238 eligible patients. These patients will be randomly assigned in a 1:1 ratio to receive either sivelestat sodium or placebo via continuous intravenous infusion (0.2mg/kg/h) over a 24-hour period for 7 days (or to the day of death or ICU discharge if it occurs before day 7). Both the patients and investigators are blinded to the treatment assignment. Subsequent follow-ups will be performed in person at 7,14 and 28 days after randomization. The primary endpoint will be at 7 days post randomization and secondary endpoints will be at 14 and 28 days post randomization. Also, endpoint assessors are masked to the treatment allocation. Lastly, these endpoint variables will be compared between the treatment groups to investigate the efficacy and safety of sivelestat for COVID-19-associated ARDS

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Confirmed SARS-CoV-2 infection as determined by Polymerase Chain Reaction (PCR) in sputum, nasopharyngeal swabs, or oropharyngeal swabs
* Diagnosis of acute respiratory distress syndrome (ARDS) according to the Berlin Definition criteria
* Onset of ARDS less than 72 hours before randomization
* Written informed consent

Exclusion Criteria:

* ARDS potentially caused by extra-pulmonary reasons, including non-pulmonary sepsis, pancreatitis, multiple trauma and massive transfusion, etc.
* Leukopenia (leukocyte count <4,000/μL/) and/or thrombocytopenia (platelet count <100,000/μL)
* Significant hepatic dysfunction, defined as elevated AST and ALT ≥ 3 times the normal limits, or total bilirubin ≥ 1.5 mg/dL
* Severe renal insufficiency with serum creatinine > 3.0 mg/dL
* History of moderate to severe chronic lung disease requiring home-based oxygen therapy, including chronic obstructive pulmonary disease (COPD), interstitial lung disease (ILD), asthma and bronchiectasis, etc.
* Pre-existing peripheral nerve injury, spinal cord trauma, or neuromuscular disorder that may impair spontaneous ventilation (e.g., high cervical spinal cord injury, Guillain-Barré Syndrome, and myasthenia gravis, etc.)
* Current diagnosis of pulmonary embolism
* Coexisting multi-organ failure, affecting more than 3 systems
* Combined with burn injury
* Life expectancy less than 6 months (e.g., due to an an end-stage malignant disease)
* Moribund and expected to die within 48 hours
* Known allergy to sivelestat or any of the study drug excipients
* Pregnancy or lactation, or the possibility of conception
* Current or recent (last 3 months) participation in any other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2023-01-31 (Estimated); Primary Completion 2024-01-03 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio | From randomization to day 7
  Changes in the PaO2/FiO2 ratio

SECONDARY OUTCOMES:
Ventilator-Free days | From randomization to day 28
  The number of Ventilator-Free Days
In-hospital mortality | Through study completion, a period of 28 days
  The rate of death during hospitalization
Length of hospitalization | Through study completion, a period of 28 days
  The overall length of hospital stay
Intensive care unit (ICU) length of stay | Through study completion, a period of 28 days
  The time interval between ICU admission and ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Guangzhi Shi, M.D., Principal Investigator — Department of Critical Care Medicine, Beijing Tiantan Hospital, Capital Medical University; Zhigang Zhao, M.D., Principal Investigator — Department of Pharmacy, Beijing Tiantan Hospital, Capital Medical University

IPD SHARING:
Plan to Share IPD: No